CLINICAL TRIAL: NCT04527822
Title: Effect of Discharge Planning Program on Patient's Outcomes Post Coronary Artery Bypass Graft Surgery
Brief Title: Discharge Planning Program for Post CABG Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Jordanian Royal Medical Services (Other)
Responsible Party: Principal Investigator, Jafar Alshraideh, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 101271-2
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Bypass Graft Surgery; Mace; 30 Day Mortality
Keywords: Coronary artery bypass graft surgery CABGl; MACE; nursing care

STUDY DESIGN:
Intervention Model Description: 2 groups Post test only
Masking Description: Non pharmacological intervention with no blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discharge planning program (Experimental): a discharge planning program. It is a modified discharge planning program depends basically on the Re-Engineered Discharge program which is a program developed by Boston Medical Center in collaboration with AHRQ , 2013. The intervention consists of several components. The program components include making appointments for follow-up care (e.g., medical appointments and post discharge tests/labs). Plan for the follow-up of results from tests or labs that are pending at discharge. Identify the correct medicines and a plan for the patient to obtain them. Teach a written discharge plan the patient can understand. Educate the patient about his or her diagnosis and medicines. Review with the patient what to do if a problem arises. Assess the degree of the patient's understanding of the discharge plan and provide a telephone reinforcement of the discharge plan
  Interventions: Other: Nurse led discharge planning program
- Standard Care (Active Comparator)
  Interventions: Other: Nurse led discharge planning program

INTERVENTIONS:
Other: Nurse led discharge planning program — a discharge planning program. It is a modified discharge planning program depends basically on the Re-Engineered Discharge program which is a program developed by Boston Medical Center in collaboration with AHRQ , 2013. The intervention consists of several components. The program components include making appointments for follow-up care (e.g., medical appointments and post discharge tests/labs). Plan for the follow-up of results from tests or labs that are pending at discharge. Identify the correct medicines and a plan for the patient to obtain them. Teach a written discharge plan the patient can understand. Educate the patient about his or her diagnosis and medicines. Review with the patient what to do if a problem arises. Assess the degree of the patient's understanding of the discharge plan and provide a telephone reinforcement of the discharge plan

SUMMARY:
The current study is utilizing a nurse led discharge program based on the Re-Engineered Discharge program (Project-RED) ( Agency of Healthcare Research and Quality [AHRQ], 2013) which is a package of services designed to minimize discharge failures and minimize re-admissions, reduce mortality, morbidity, complication and improve patients outcomes. Project-RED aims to reduce hospital re-admissions through a series of structured steps led by a nurse called discharge advocate. The intervention will be used to discharge patients post Coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the main threats to human lives (Benjamin et al., 2018). Around 17.9 million deaths worldwide were attributed to CVD (Benjamin et al., 2018); Which Represents 31 % of the global deaths (Benjamin et al., 2018). Coronary artery disease is one of the CVD. Coronary artery disease prevalence among United State (US) adults aged 20 years and above is 6.3 %. It is responsible for 43.8 % of the deaths worldwide. (Benjamin et al., 2018).

In Jordan, CVD is the leading cause of death. During 2016; 37 % of all deaths among Jordanian population were due to CVD. Coronary Artery Disease is responsible for 18 % of the deaths (Centers of Disease Control [CDC], 2016) Coronary artery diseases currently are managed with medical treatment, percutaneous coronary interventions (PCI) or Coronary artery bypass graft (CABG) surgery (Habib et al., 2015). Coronary artery bypass graft surgery is the indicated choice for multi-vessel coronary disease (Habib et al., 2015). It is defined as a revascularization procedure used for the treatment of CAD. It involves establishing a graft from another vessel of the body to bypass the narrowed coronary artery and restore blood flow to the cardiac muscle (Urden, Stacy, & Lough, 2017).

Even though Coronary Artery Bypass Graft surgery is believed to provide more complete revascularization and leading to improved long term outcomes than PCI (Hillis et al., 2011); the recovery process after hospital discharge might be complicated by the occurrence of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) (Goldfarb et al., 2015). Major Adverse Cardiovascular and Cerebrovascular Events consist of mortality, myocardial infarction (MI), stroke and need for repeat revascularization (Goldfarb et al., 2015). Mortality leads to losing the patient after a major and costly surgery, while; MI, stroke and need for reopening or repeat revascularization leads to patient readmission to the hospital and might end up with increased mortality rate (Goldfarb et al., 2015; Hillis et al., 2011).

Mortality rate after CABG ranges from 1.1% -24 % (Grundeken et al., 2013; Jose et al., 2019; Shah et al., 2019; Wrobel et al., 2015). Among the Jordanian CABG population; all-cause mortality reported 30 day after surgery was 5.9 % in 1046 patients (AlWaqfi, Khader, & Ibrahim, 2012).

The readmission rate of CABG patients within 30 days is seriously high (Feng, White, Gaber-Baylis, Turnbull, & Rong, 2018). More specifically; Feng et al., (2018) reported that 28601 adult CABG patients out of 177229 (16 %) in the united States (US) were readmitted within 30 days (Feng et al., 2018). Another study revealed that more than 60 % of CABG patients readmissions occur within the first week post discharge (Price, Romeiser, Gnerre, Shroyer, & Rosengart, 2013). Several reasons stand behind hospital readmissions after CABG surgery (Mary, 2017; Seifert, 2017). Price et al., (2013) reported that 25% of 13% hospital readmissions after CABG surgery were attributed to cardiac reasons.

Myocardial Infarction after CABG surgery is Type 5 MI (Thygesen et al., 2018). Shah et al., (2016) reported that out of 2215 CABG patients 5.8 % developed acute MI post-surgery while 3.8 % required repeat revascularization. Repeat revascularization is a new CABG or PCI procedure needs to be done due to documented ischemia or graft failure and it is one of the MACCE that might occur within 30 days after CABG surgery (Takagi et al., 2013). The incidence rate of repeated revascularization among CABG patient is ranging from 0.5 % -1.3 % (Deppe et al., 2016; Taggart et al., 2015; Wu et al., 2015) Stroke is an acute focal neurological deficit lasting ≥ 24 hours with or without confirmatory imaging (Goldfarb et al., 2015). Around 1.3% of CABG patients developed stroke after the surgery which causes near 20 % mortality rate perioperative (Gaudino et al., 2019). Among Jordanian population; CABG Patients who had stroke were 2.3 % of the sample (1046 patients). Of these; 33.3 % were died (AlWaqfi et al., 2012).

Reducing mortality and hospital readmission following cardiac surgery has become a national priority in the US and worldwide. Unclear discharge instructions and lack of follow up plans are among the reported reasons for hospital readmissions (Amoah & Mwanri, 2016). Patient experience with discharge instructions show that patients who discharged with sufficient information and provided follow-up care were better in managing postoperative problems and experienced improved post discharge outcomes (M. Akbari & Celik, 2015). Therefore; have a better health-related quality of life (HRQOL).

The current study intervention is a nurse led discharge program based on the Re-Engineered Discharge program (Project-RED) ( Agency of Healthcare Research and Quality [AHRQ], 2013) which is a package of services designed to minimize discharge failures and minimize readmissions (Jack et al., 2009; S. Mitchell, Weigel, Laurens, Martin, & Jack, 2017; S. E. Mitchell et al., 2016; Patel & Dickerson, 2018), reduce mortality, morbidity, complication (Ceppa et al., 2015) and improve patients outcomes (Adams, Stephens, Whiteman, Kersteen, & Katruska, 2014; Berkowitz et al., 2013; Cancino et al., 2017) . Project-RED aims to reduce hospital readmissions through a series of structured steps led by a nurse called discharge advocate. (Jack et al., 2009)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 21 years or older
* Underwent first time isolated elective CABG surgery for single, double, or triple CAD.
* Patient speak and read Arabic to eliminate any barriers of communication during the process of discharge and telephone call
* Patient who has contact telephone number
* Doesn't have Aortic calcification, and /or previous stroke
* Welling to participate and Able to provide informed consent

Exclusion Criteria:

* Adult patient aged 21 years or older
* Underwent first time isolated elective CABG surgery for single, double, or triple CAD.
* Patient speak and read Arabic to eliminate any barriers of communication during the process of discharge and telephone call
* Patient who has contact telephone number
* Doesn't have Aortic calcification, and /or previous stroke
* Welling to participate and Able to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | 30 days
  The variable of MACCE includes MI, Stroke, and all-cause death and repeat re-vascularization

SECONDARY OUTCOMES:
Adherence to medications | 3 months
  Adherence to medications

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No